CLINICAL TRIAL: NCT02307890
Title: The Relationship of Hepatobiliary microRNA Expression Profile and Clinical Outcome in Liver Transplantation
Brief Title: The Relationship of Initial Liver Profile and Outcome After Transplantation
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2014/097
Record Dates: First submitted 2014-11-24; First posted 2014-12-04 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Liver Failure
Keywords: Liver Transplantation
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver and bile duct
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver transplantation group: Participants will include all deceased adult liver transplant donors (>16 years of age) whose livers are being utilised for transplantation in the Scottish Liver Transplant Unit in the Royal Infirmary of Edinburgh. Exclusion criteria will include paediatric liver transplant donors (<16 years of age).

SUMMARY:
Donation after cardiac death (DCD) livers are increasingly utilised in liver transplantation but concerns exist regarding negative results. Ischemic cholangiopathy (IC) is damage to one or more bile ducts probably caused by inadequate blood flow or a failure of biliary epithelium to regenerate. It typically presents weeks to months after liver transplantation, is often refractory to treatment and can result in a requirement for re-transplantation. Although IC is more common following DCD liver transplantation, it is otherwise very difficult to predict and the underlying pathogenesis is poorly understood. The aim of this study is to correlate microRNA (miRNA) levels and markers of senescence in liver and bile duct biopsies taken during liver transplantation with the incidence of IC following liver transplantation.

DETAILED DESCRIPTION:
Study population

Tissue from all deceased adult liver transplant grafts will be collected. The test samples will be selected from procedures were the liver transplant recipient has developed IC. The control samples will include tissues from procedures were the transplant recipient had an uncomplicated outcome. There will be matching of test samples and control samples based on a range of clinical factors.

Consent

Standard consent for organ donation documentation has a general consent to research section. Due to the small risk of damage to blood vessels when taking samples the liver transplant recipient will also be consented for these procedures to take place.

Tissue sampling

Liver and bile duct samples from each graft will be obtained at various different time points during liver transplant procedures.

Processing of specimens

Following removal of the specimens, samples will be divided then added to RNAlater (Life Technologies, Paisley, UK), 10% formaldehyde or will be snap frozen. At a later time point samples will be analysed.

Definition of ischemic cholangiopathy

IC will be defined as strictures, dilatations, or irregularities of the intra- or extrahepatic bile ducts of the liver graft. Isolated strictures at the bile duct anastomosis will be excluded. The diagnosis will be based on at least one adequate imaging study of the biliary tree, after exclusion of hepatic artery thrombosis by Doppler ultrasound, computed tomography or conventional angiography.

ELIGIBILITY:
Inclusion Criteria:

* All deceased adult liver transplant donors (>16 years of age) whose livers are being utilised for transplantation in the Scottish Liver Transplant Unit in the Royal Infirmary of Edinburgh

Exclusion Criteria:

* Paediatric liver transplant donors (<16 years of age).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Liver transplantation group
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-08-06 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in hepatobiliary miRNA expression during liver transplantation in liver grafts that develop ischemic cholangiopathy following liver transplantation | 12 months
  Assessed by sequencing of liver and bile duct samples taken during different stages of liver transplantation and correlation with clinical outcomes

SECONDARY OUTCOMES:
Changes in hepatobiliary senescence during liver transplantation in liver grafts that develop ischemic cholangiopathy following liver transplantation | 12 months
  Assessed by senescence markers in liver and bile duct samples taken during different stages of liver transplantation and correlation with clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Ewen Harrison, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Neill S, Roebuck A, Khoo E, Wigmore SJ, Harrison EM. A meta-analysis and meta-regression of outcomes including biliary complications in donation after cardiac death liver transplantation. Transpl Int. 2014 Nov;27(11):1159-74. doi: 10.1111/tri.12403. PMID 25052036